CLINICAL TRIAL: NCT00950365
Title: A Randomized Phase II Study of Schedule-Modulated Concomitant Pemetrexed (Alimta) and Erlotinib (Tarceva) vs Single Agent Pemetrexed (Alimta®) in Patients With Progressive or Recurrent Non-small Cell Lung Cancer (NSCLC)
Brief Title: Pemetrexed Disodium With or Without Erlotinib Hydrochloride in Treating Patients With Stage IIIB-IV or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eli Lilly and Company (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Roman Perez-Soler, Principal Investigator, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-10-277; NCI-2013-01128 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 05277; 05-10-277 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Bronchioloalveolar Carcinoma; Large Cell Lung Carcinoma; Lung Adenocarcinoma; Recurrent Non-Small Cell Lung Carcinoma; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma, Bronchiolo-Alveolar; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (pemetrexed) (Active Comparator): Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium
- Arm B (pemetrexed disodium, erlotinib hydrochloride) (Experimental): Patients receive pemetrexed disodium IV as in Arm A and erlotinib hydrochloride PO QD on days 2-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
  Arms: Arm B (pemetrexed disodium, erlotinib hydrochloride)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt

SUMMARY:
This randomized phase II trial studies how well pemetrexed disodium with or without erlotinib hydrochloride works in treating patients with stage IIIB-IV or recurrent non-small cell lung cancer. Drugs used in chemotherapy, such as pemetrexed disodium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether pemetrexed disodium is more effective with or without erlotinib hydrochloride in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate progression free survival (PFS) in the schedule-modulated concomitant administration of erlotinib (erlotinib hydrochloride) and pemetrexed (pemetrexed disodium), and in single agent pemetrexed in patients with advanced non-small cell lung cancer (NSCLC) as second-line chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate antitumor objective response rate (complete response [CR] + partial response [PR]) per Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

II. To evaluate disease control rate (response rate + stable disease, i.e., CR+PR+ stable disease [SD]) and duration of response.

III. To evaluate median time to progression (TTP) and overall survival (OS). IV. To evaluate the safety profile of concurrent pemetrexed and erlotinib versus single agent pemetrexed.

TERTIARY OBJECTIVES:

i. To determine several molecular and cellular biomarkers in the tumors, the skin and the serum that are predictive of the efficacy of pemetrexed and erlotinib.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive pemetrexed disodium intravenously (IV) over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive pemetrexed disodium IV as in Arm A and erlotinib hydrochloride orally (PO) once daily (QD) on days 2-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced (stage IIIB with a malignant pleural effusion or stage IV disease) or recurrent nonsquamous NSCLC
* Patients must have at least one measurable disease per RECIST criteria; all sites of disease must be assessed within 4 weeks prior to registration
* Patient must have disease progression after one prior combinational chemotherapy and/or targeted therapy other than pemetrexed or an epidermal growth factor receptor (EGFR) ) tyrosine kinase inhibitor (TKI) (such as erlotinib, gefitinib, or a second generation EGFR TKI); prior monoclonal antibody against EGFR is allowed) for metastatic disease, or relapse while receiving adjuvant therapy, or within 12 months of completing adjuvant therapy
* All patients will be screened for brain metastasis within 6 weeks prior to registration; patients with treated and stable brain metastases must have been treated with surgery and/or radiation and are asymptomatic and are no longer taking corticosteroids
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 or Karnofsky >= 60%
* Absolute neutrophil count >= 1,500/uL
* Hemoglobin >= 8.0 g/dL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN), except in known hepatic metastasis, wherein may be =< 3.0 X ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN, except in known hepatic metastasis, wherein may be =< 5.0 X ULN
* Creatinine clearance >= 45 mL/min for patients with creatinine levels above institutional normal
* Patients must not be pregnant or breastfeeding since there is no information regarding the use of these agents in this population; a negative serum or urine pregnancy test is required within 14 days prior to registration if pre- or perimenopausal (i.e., last menstrual period within one year of registration); both pemetrexed and erlotinib are Class D agent with the potential for teratogenic or abortifacient effects; patients both females and males with reproductive potential (i.e. menopausal for less than 1 year and not surgically sterilized) must practice contraceptive measures throughout the study
* Patients taking Warfarin or nonsteroidal anti-inflammatory drugs (NSAIDs) are eligible; patients with mild to moderate renal insufficiency should avoid taking NSAIDs with short elimination half-lives for a period of 2 days before, the day of, and 2 days following administration of Alimta; if the patient is taking other cytochrome P450 3A4 (CYP3A4) inducers or inhibitors, they must be discontinued at least one week prior to starting erlotinib
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had immunotherapy, hormone, chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have received pemetrexed or an EGFR TKI (such as erlotinib, gefitinib, or a second generation anti-EGFR TKI) for their metastatic disease should be excluded from this clinical trial; other molecularly targeted agent, including monoclonal antibody or vaccine against EGFR or angiogenesis inhibitor, is allowed
* Patients may not be receiving any other investigational or commercial agents or therapies other than those described below with the intent to treat the patient's malignancy
* Patients with uncontrolled brain metastases should be excluded from this clinical trial because of their poor prognosis
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib or pemetrexed or other agents used in the study
* Patients with gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease, are ineligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (such as bacteremia or active hepatitis), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with erlotinib or pemetrexed or other agents administered during the study; appropriate studies will be undertake in patients receiving combination anti-retroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2006-04; Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Perez-Soler, Principal Investigator — Albert Einstein College of Medicine
Locations (5):
- United States (5):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - Albert Einstein College of Medicine, The Bronx, New York
  - Bronx River Medical Associates PC, The Bronx, New York
  - Eastchester Center for Cancer Care, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with platinum-treated metastatic non squamous NSCLC randomly assigned 1:2 to pemetrexed alone (500 mg/m^2 provided iv on day 1) or pemetrexed followed by erlotinib (150 mg provided orally daily on days 2-17) every 21 days.
Period: Overall Study
Arm/Group | Arm A (Pemetrexed) | Arm B (Pemetrexed Disodium, Erlotinib Hydrochloride)
Started | 27 | 52
Completed | 25 | 50
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Pemetrexed) | Arm B (Pemetrexed Disodium, Erlotinib Hydrochloride) | Total
Number analyzed (Participants) | 27 | 52 | 79
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [47 to 91] | 62 [37 to 86] | 63 [37 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 29 | 42
  Male | 14 | 23 | 37
Race/Ethnicity, Customized [Number; unit: participants]
  White | 18 | 36 | 54
  Black | 5 | 9 | 14
  Hispanic | 4 | 6 | 10
  Asian | 0 | 2 | 2
Smoking history [Number; unit: participants]
  <=15 pack-years | 5 | 17 | 22
  >15 pack-years | 22 | 35 | 58
ECOG PS [Number; unit: participants] — ECOG PERFORMANCE STATUS:
  0- Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities
  participants
    ECOG PS 0 | 24 | 46 | 70
    ECOG PS 1/2 | 3 | 6 | 9
Histology: Nonsquamous [Number; unit: participants]
  Prior platinum-containing chemotherapy | 27 | 50 | 77
  Prior antiangiogenic inhibitor | 10 | 18 | 28
Evaluable patients with atleast one source of biospecimen [Number; unit: participants]
  Archival tumor specimens | 6 | 14 | 20
  Collected blood samples | 17 | 32 | 49
  EGFR (epidermal growth factor receptor) wild type | 21 | 31 | 52
  EGFR (epidermal growth factor receptor) mutations | 0 | 7 | 7
  Unkown EGFR (epidermal growth factor recep) status | 4 | 12 | 16

OUTCOME MEASURES:

1. Primary Outcome: PFS (Progression Free Survival)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Time from randomization until documented tumor progression or death from any cause, assessed up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Pemetrexed) | Arm B (Pemetrexed Disodium, Erlotinib Hydrochloride)
Number analyzed (Participants) | 25 | 50
months | 8 [0 to 19] | 20 [7 to 29]

2. Secondary Outcome: Objective Response Rate (CR +PR) Evaluated Using RECIST
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
  Response rates in each arm will be summarized by computing proportions and corresponding 95% confidence intervals.
Time Frame: Up to 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Pemetrexed) | Arm B (Pemetrexed Disodium, Erlotinib Hydrochloride)
Number analyzed (Participants) | 25 | 50
percentage of participants | 12 [0 to 25] | 28 [10 to 40]

3. Secondary Outcome: Overall Survival
Description: Time to event endpoints will be analyzed using standard survival analytic methods, including the Kaplan-Meier approach for estimating the survival distributions.
Time Frame: Time from the date of randomization to date of death due to any cause, assessed up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Pemetrexed) | Arm B (Pemetrexed Disodium, Erlotinib Hydrochloride)
Number analyzed (Participants) | 25 | 50
Participants | 25 | 50

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm A (Pemetrexed) | Arm B (Pemetrexed Disodium, Erlotinib Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/50
Serious Adverse Events (participants affected / at risk) | 9/25 | 16/50
Other Adverse Events (participants affected / at risk) | 25/25 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Pemetrexed) (N=25) | Arm B (Pemetrexed Disodium, Erlotinib Hydrochloride) (N=50)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 10 (10)
Insterstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Pemetrexed) (N=25) | Arm B (Pemetrexed Disodium, Erlotinib Hydrochloride) (N=50)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 17 (17)
Nausea (Gastrointestinal disorders) | 4 (4) | 20 (20)
Vomiting (Gastrointestinal disorders) | 2 (2) | 13 (13)
Mucositis (Gastrointestinal disorders) | 0 (0) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 23 (23)
Dehydration (General disorders) | 3 (3) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 13 (13)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 35 (35)
Transaminases (Endocrine disorders) | 3 (3) | 9 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5) | 15 (15)
Infection (General disorders) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 14 (14) | 33 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-04-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT00950365/Prot_SAP_000.pdf